CLINICAL TRIAL: NCT05614999
Title: The Validation and Efficacy of Varix Trainer as a Training Device Esophagogastroduodenoscopy (a Multicenter Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3741
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Gastric Varix
Keywords: Endoscopy training, Gastroscopy, Tip control, Motor skill
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): Participants in this group will do the pre-training test, practicing eight-sessions (each session is approximately 15minutes) and then do the post-training test.
  Interventions: Other: Endoscopy training curriculum
- Non-training group (No Intervention): Participants in this group will do the pre-training test, and then do the post-training test after the pre-test 4-6weeks.

INTERVENTIONS:
Other: Endoscopy training curriculum — Eight sessions training in endoscopic tip control using Varix trainer model I.
  Arms: Training group

SUMMARY:
The goal of this exploratory validation study is to compare levels of expertise (or non-expertise) between GI fellows and experts with the varix trainer. The main question it aim to answer is:

Can the varix trainer distinguish levels of expertise (or non-expertise) between novices and experts for specific skills (torque, small wheel and retroflexion techniques)? Does the training with the varix trainer improves these specific skills of GI fellows? Participants will do the pre-training test, practicing eight-sessions (each session is approximately 15minutes) and then do the post-training test.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled participants from Ramathibodi hospital King Chulalongkorn Memorial hospital Siriraj hospital Rajavithi hospital Vajira hospital Nanthana-Kriangkrai Chotiwattanaphan Institute of Gastroenterology and Hepatology Srinagarind Hospital

  1. Expert (> 1,500 EGD)
  2. Trainees (First and second year fellow)

Exclusion Criteria:

* Deny to participate in our study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-06 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Motor skill for endoscopic tip control improvement VS control | 4-6 weeks
  Speed of pointing to 20 numbers using Varix trainer model I

SECONDARY OUTCOMES:
Motor skill for endoscopic tip control 1st year fellow trainee VS 2nd year fellow trainee VS expert | 4-6 weeks
  Speed of pointing to 20 numbers using Varix trainer model I

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No